CLINICAL TRIAL: NCT00754481
Title: Hypothermia for Cardiac Arrest in Paediatrics (HypCAP) - Pilot Study
Brief Title: Hypothermia for Cardiac Arrest in Paediatrics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jamie Hutchison, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000004888
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Arrest
Keywords: Paediatrics
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Other: Normothermia
- 2 (Experimental)
  Interventions: Other: Hypothermia

INTERVENTIONS:
Other: Normothermia — Patients randomized to the Normothermia arm (esophageal temp 36.5-37.5 ºC) were maintained at an esophageal temperature of 36.5-37.5ºC for 48 hours. Patients who were hypothermic (temperature < 35 ºC) when randomized to the normothermia group were rewarmed slowly using the servo-controlled mattress. Patients who were hyperthermic following randomization to the normothermia group were actively cooled to normothermia using the servo-controlled mattress. Neuromuscular blockers were administered as needed intravenously in both groups of patients to prevent shivering.
  Arms: 1
Other: Hypothermia — Patients randomized to the Hypothermia arm (esophageal temp 33º to 34 °C) were cooled rapidly using the cooling protocol developed for the Hypothermia Paediatric Head Injury Trial. A temperature probe was placed in the esophagus and its position confirmed using a chest radiograph. Patients were placed on a servo-controlled cooling blanket and covered in crushed ice (in sealed plastic bags covered by pillow cases) and a second cooling blanket. Once the esophageal temperature reached 34.0ºC, the ice and second cooling blanket was removed and esophageal temperature was maintained at 33º to 34 °C for 48 hours using the servo-controlled cooling mattress. Patients treated with ECMO were cooled using the extracorporeal circuit cooling-device. Rewarming was done at a rate of 0.5 ºC every 2 hours until an esophageal temperature of 36.5 ºC was reached. Thereafter temperature was recorded but not controlled by surface cooling.
  Arms: 2

SUMMARY:
The investigators hypothesized that, following cardiac arrest in pediatric patients, hypothermia therapy will improve the proportion of patients with a good functional outcome compared to a normothermic control group.

DETAILED DESCRIPTION:
Cardiac arrest is associated with a high morbidity and mortality in children and hypothermia therapy has the potential to be beneficial in children following cardiac arrest. We have a track record of both clinical and laboratory research of hypothermia therapy following cardiac arrest at the Hospital for Sick Children and have completed a 3-site randomized controlled pilot study of hypothermia therapy following cardiac arrest in children funded by The Hospital for Sick Children Research Institute and the Heart and Stroke Foundation of Ontario. This protocol was used to develop the protocol for the THAPCA trials (see 2 manuscripts published Moler et al NEJM 2015 and 2017 and multiple other manuscripts). Hypothermia therapy, compared to active maintenance of normothermia, had no beneficial effect on functional outcome or mortality in children with out-of-hospital or in-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by parent or legal guardian
* Age ≥ 38 weeks gestation up to and including 17 years
* Patient admitted with a diagnosis of a cardiac arrest requiring compressions ≥3 minutes
* Remain comatose i.e. have Glasgow Coma Score less than or equal to 10 assessed at the tertiary level pediatric hospital at least 1 hour post- cardiac arrest
* Invasive mechanical ventilation

Exclusion Criteria:

* Cardiac arrest lasting ≥45 minutes, irregardless of commencement of ECMO
* Refractory hemorrhagic shock
* Dysrhythmia leading to cardiac arrest, where cooling would be part of standard therapy
* Suspected diagnosis of brain death as defined as fixed and dilated pupils, Glasgow Coma Score of 3 and no evidence of brain function on neurological examination
* Patients who have had a prolonged cardiac arrest at the scene of a trauma
* Decision to withhold (DNR) or withdraw life sustaining therapies
* Acute Birth asphyxia
* Terminal illness, not expected to survive 12 months
* Cardiac arrest caused by septic shock
* Severe neurodevelopmental disability or persistent vegetative state prior to cardiac arrest
* Near drowning in ice water and temperature <32ºC on admission to study site
* It has been more than 6 hours following cardiac arrest (estimated by first responder)
* Previous enrolment in the HypCAP Pilot Study
* Pregnant
* Parent/Guardian refuse consent
* Responsible physician refuses to enrol patient

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2005-01; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The percentage of children achieving a "good outcome", that is, a PCPC of 1-3 will be assessed using the Paediatric Cerebral Performance Category scores | Assessed at 12 months post cardiac arrest

SECONDARY OUTCOMES:
Cognitive and motor measures | Assessed at 12 months post-arrest
Mortality | Assessed at 1, 3, 6, and 12 months post-arrest
Cerebral edema | 12 months
Adverse effects of hypothermia therapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Hutchison, MD, Principal Investigator — The Hospital for Sick Children
Locations (4):
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Sainte-Justine Hospital, Montreal, Quebec
- Starship Children's Hospital, Auckland, New Zealand
- Great Ormond Street Hospital, London, United Kingdom